CLINICAL TRIAL: NCT03113084
Title: Phase I Study With Pharmacodynamic Determination of Unfractionated Heparin of Porcine Origin of the Company União Química of Subcutaneous Use in Healthy Participants
Brief Title: Study With Heparin Sodium in Subcutaneous Administration
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Delay in the R&D stage
Sponsor: União Química Farmacêutica Nacional S/A (Industry)
Collaborators: Buranello e Rodrigues Consultoria em Desenvolvimento Farmacêutico Ltda ME (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PGUQ003
Record Dates: First submitted 2017-03-29; First posted 2017-04-13 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-06

CONDITIONS: Heparin
Keywords: Sodium Heparin; Pharmacokinetics; Coagulation factor

STUDY DESIGN:
Intervention Model Description: Hospitalizations for administration of study medications will occur in two periods (visits 1 and 2) for administration of the drugs, and participants who receive the test medication at visit 1 will receive the comparator medication at Visit 2 and vice versa.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group Sodium Heparin UQ First (Experimental): The participants will receive the Sodium heparin UQ subcutaneous drug administration at first period and the Sodium heparin FK subcutaneous drug administration at second period
  Interventions: Biological: Sodium Heparin UQ subcutaneous drug administration; Biological: Sodium Heparin FK subcutaneous drug administration
- Group Sodium Heparin FK First (Experimental): The participants will receive the Sodium heparin FK subcutaneous drug administration at first period and the Sodium heparin UQ subcutaneous drug administration at second period
  Interventions: Biological: Sodium Heparin UQ subcutaneous drug administration; Biological: Sodium Heparin FK subcutaneous drug administration

INTERVENTIONS:
Biological: Sodium Heparin UQ subcutaneous drug administration — The participants will be hospitalized one day to receive the Sodium heparin UQ experimental medication or Sodium heparin FK comparator medication. They will receive the Subcutaneous medication and start the blood collection at the programmed time. After 7 days, the participants will return to receive the other medication and have their blood collected. The last visit will be to collect safety datas
Biological: Sodium Heparin FK subcutaneous drug administration — The participants will be hospitalized one day to receive the Sodium heparin FK comparator medication or Sodium heparin UQ experimental medication. They will receive the subcutaneous medication and start the blood collection at the programmed time. After 7 days, the participants will return to receive the other medication and have their blood collected. The last visit will be to collect safety datas

SUMMARY:
The purpose of this phase I study is to know the pharmacodynamic profile in humans of the sodium heparin of porcine origin of the company União Química, building from the pharmacodynamic data generated its pharmacokinetic profile, due to the dosage limitation of heparin directly in biological samples. In addition, the toxicity of the product will be evaluated in healthy male participants.

DETAILED DESCRIPTION:
This stage of product development follows the guidelines of the ANVISA (National Health Surveillance Agency) Heparin Development Guide.

Unfractionated sodium heparin is a drug known and widely used in the world for over half a century, thus, no unknown adverse events or any risk of administration are expected in humans, however, this is the first human Biological product developed by União Química. The proposed development of this biological drug follows the individual route, the control heparin used in the present study has the objective of evaluating the results found with the test product, without the obligation to demonstrate bioequivalence among the evaluated products.

ELIGIBILITY:
Inclusion Criteria:

* Eligible healthy participants should sign the Informed Consent Form,
* be between 18 and 60 years of age,
* be male,
* present a BMI ≥ 18.5 and ≤ 29.9 kg / m2,
* be characterized as a voluntary (Normal physical examination)
* no history of current or recent diseases.

Exclusion criteria:

* hemoglobin <12 g / dL;
* Platelets <100 x 109 / L;
* Regular or last 30 days use of anticoagulant medications;
* Current or past use of anti-inflammatory or anti-platelet medications;
* History of gastrointestinal bleeding;
* History of venous thrombosis, pulmonary embolism, coagulopathies or any coagulation disorder;
* Any other chronic illness or regular use of drugs that at the discretion of the investigator contraindicates participation in the study,
* serious comorbidity (at the discretion of the researcher) of any nature that could compromise participation in the study or put the participant at risk considered to be unacceptable,
* Laboratory that at the discretion of the investigator contraindicates the participation of the participant in the study;
* Hypersensitivity or contraindication to the components of the medications studied, participation in another clinical study in less than 1 year (unless justified by the investigator)
* donation of blood (> 500 mL) in the preceding 3 months.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — It is known that male participants are preferable in clinical trials due to the hormonal stability presented by males compared to females, and the results that the drug under test can present are clearer, that is, with less hormonal interference.
Enrollment: 38 (Estimated)
Dates: Start 2022-08-20 (Estimated); Primary Completion 2023-04-20 (Estimated); Study Completion 2023-10-10 (Estimated)

PRIMARY OUTCOMES:
Activity of the anti-Xa factor | 8 hours
  Chromogenic determination of direct and indirect inhibitors in human citrated plasma

SECONDARY OUTCOMES:
Activity of anti-IIa factor | 8 hours
  Chromogenic determination of direct and indirect inhibitors in human citrated plasma
activity of anti-Xa / anti-IIa ratio | 8 hours
  the calculated ratio of the activity of anti-Xa / anti-IIa
activity of tissue factor pathway activity (TFPI) | 8 hours
  the Elisa assay will determine the activity of tissue factor pathway activity (TFPI)
adverse events | 45 days
  Adverse events occurred in the study

CONTACTS AND LOCATIONS:
Overall Officials: Paula F Santos, Study Director — União Química Farmacêutica Nacional S/A
Locations (1):
- União Química Farmacêutica Nacional, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No